CLINICAL TRIAL: NCT05285150
Title: Weighting of Balance Deficiencies Performed by Physical Therapist in Argentina in Subjects With Risk of Falling
Brief Title: The Weighting of the Balance
Status: Completed | Type: Observational
Sponsor: Hospital de Rehabilitacion Manuel Rocca (Other)
Responsible Party: Principal Investigator, Gerardo Candoni, Physical Therapy, Hospital de Rehabilitacion Manuel Rocca
Other Study IDs: 6550
Record Dates: First submitted 2022-03-04; First posted 2022-03-17 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Physical Therapy; Survey; Balance; Assessment
Keywords: Physical Therapy; Survey; Balance; Assessment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — It´s a survey

SUMMARY:
Summary Introduction: Falls are involuntary events that cause loss of balance and hit the body on the ground or on another firm surface that stops it. 40% of people with various neurological disorders fall one or more times, and of all these, 21% suffer a fall-related injury. Objective and instrumented gait analysis is an important tool for estimating the risk of falls in patients.

Objective: To describe the protocols used by physical therapist residing in Argentina when categorizing a balance problem within the framework of neurorehabilitation, vestibular rehabilitation, geriatrics and gerontology. Identify the barriers and facilitators self-perceived by physical therapist that make it difficult to weight deficiencies in balance.

Method: An observational, descriptive, cross-sectional study of the online survey type will be carried out. The recommendations given by the Checklist for Reporting of Survey Studies will be used. The survey, which was created by the researchers of this study, will consist of 26 items divided into 4 sections. It will be aimed at all those physical therapist in Argentina who are dedicated to neurorehabilitation, vestibular rehabilitation, geriatrics and gerontology. The type of sampling used will be non-probabilistic by snowball, which will be done online through the SurveyMonkeyTM tool.

DETAILED DESCRIPTION:
Materials and method Study design An observational, descriptive, cross-sectional study will be carried out. For its future report, the recommendations given by the Checklist for Reporting of Survey Studies (CROSS) will be used.

Sample Characteristics All those physical therapist and related degrees dedicated to neurorehabilitation/vestibular rehabilitation/geriatrics and gerontology who practice in Argentina and who have experience in weighing balance deficiencies in subjects at risk of falling will be included. All surveys with missing data will be excluded. The type of sampling used will be non-probabilistic by snowball.

Data collection methods The online type survey which was created by the researchers of this study, will be made up of 25 items divided into 4 sections, a restriction will be created in each item to prevent respondents from leaving it without answering and those who have met all the inclusion criteria will access it.

* The first section (respondent characteristics) consists of 10 questions.
* The second section (weighting performed by the respondent) is made up of 12 questions. Those participants who choose the "no" option in question 11 will go on to the next section.
* The third section (self-perception of barriers and facilitators at the time of weighting) is made up of 2 questions.
* The fourth section (learning needs) consists of a question. Within the second section, the choice of scales was made based on a previous search in the literature about those that are most used, which to date have not been translated or adapted cross-culturally into Argentine Spanish, most of them. the same It will be aimed at all those physical therapist in Argentina who are dedicated to neurorehabilitation, vestibular rehabilitation, geriatrics and gerontology. With this purpose, a pilot test was carried out prior to the beginning of the study with the objective of the viability and understanding of the survey, it was carried out with 10 experts in the area. They were given a sheet with questions aimed at finding out the difficulties they encountered when answering the survey in general or with a particular question. Modifications were made through consensus among the authors.

Survey Administration You will be invited to participate in the study by sending the survey via email and through social network links (FacebookTM, TwitterTM, InstagramTM, LinkedinTM and WhatsappTM). The invitation will be given to specialized groups in the area, specialization careers, physical therapy colleges in the country and the Argentine association of kinesiology. The invitation will contain the objective of the study and its corresponding link to access the survey, which will be online through the SurveyMonkeyTM tool.

The period in which the current link will be maintained will be 2 months or until the required sample size is reached. To avoid multiple participation of participants, the same tool to be used (SurveyMonkeyTM) prevents double completion when using the same device. In addition, a restriction will be applied to each question, thus preventing them from leaving unanswered answers.

Sample size The required sample size will be 400 participants, since the accepted level of error will be 5%. In turn, an analysis divided by half of the consistency will be carried out, in order to determine if the results obtained are reliable or not.

Study Preparation Prior to the activation of the survey link, contact will be made throughout the previous month in different institutions and experts on the subject, with the aim of increasing the degree of knowledge and interest in it at the time of the start of the study. Contact will be made through emails and different social networks (FacebookTM, TwitterTM and InstagramTM).

Ethical considerations Given the voluntary and anonymous nature of the study, the signature of the informed consent of the participants will not be required, as established by resolution 1480/2011. Before accessing the questionnaire, participants will receive an information sheet that will include study information, investigator contact information, a privacy statement, and a statement regarding voluntary participation. At all times, the protection of the identity and data of the study participants will be preserved, in accordance with current legal regulations National Law on Protection of Personal Data 25326, in accordance with international regulations in accordance with the provisions of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapist in Argentina who are dedicated to neurorehabilitation, vestibular rehabilitation, geriatrics and gerontology.
* Practice in Argentina.
* Have experience in weighing balance deficiencies in subjects at risk of falling

Exclusion Criteria:

• All surveys with missing data will be excluded

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical therapist in Argentina who are dedicated to neurorehabilitation, vestibular rehabilitation, geriatrics and gerontology who practice in Argentina
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Balance assessment | 2022
  It will be measured through the self-report of the respondent whether or not they use a standardized scale or clinical observation with their patients. The variable will be categorized as dichotomous qualitative and the response options will be yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Rocca, Buenos Aires, Argentina